CLINICAL TRIAL: NCT06879912
Title: A Prospective, Post-Market Study to Evaluate the Clinical Utility of the Force Feedback Instruments in RAS Procedures Using the da Vinci 5 Surgical System
Brief Title: A Study to Understand the Utility of the Force Feedback Instruments in Robotic Procedures Using da Vinci 5 Robot
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dV5-MP-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hernia, Inguinal; Hernia, Ventral; Colorectal; Thoracic; Gynecologic; Partial Nephrectomy
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

SUMMARY:
The goal of this observational study is to understand the utility of force feedback instruments in surgeries that are done using the da Vinci 5 robot.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

1. Age 22 years or older
2. ASA ≤ 3
3. The clinical decision has been made to perform multi-port robotic assisted surgery with da Vinci 5 with Force Feedback instruments for the study specified procedure as primary procedure prior to enrollment in the study
4. Subject or a legally authorized representative is able to provide written informed consent using the study informed consent form prior to the study
5. Subject is willing and able to comply with the study protocol requirements including follow up schedule

Pre-operative Exclusion Criteria:

* Subject receiving an emergent procedure
* Subject planned to undergo major concomitant surgery for the treatment of a different medical condition than was originally planned
* Subject with previous ipsilateral surgery (open, endoscopic or robotic) with the same surgical indication
* Subject with past or ongoing medical conditions (for example: inflammatory bowel disease) which, in the judgment of the Investigator, puts them at high risk for surgery and not appropriate for the study
* Subject is pregnant or suspected to be pregnant or breastfeeding
* Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data
* Subject is currently participating in or has participated in a study of an investigational agent or a significant risk investigational device study within the past 6 months
* Subject belongs to a vulnerable population.
* Subject is contraindicated for anesthesia or surgery.
* Subject has had previous neoadjuvant therapy, previous chemotherapy, immunotherapy, and/or radiation therapy for the treatment of the cancer to be resected within the past 6 months

Intra-operative Exclusion Criteria

* Subject with hemodynamic or respiratory instability, which precludes the Investigator from performing the RAS.
* Subject in whom inadequate visualization makes a minimally invasive approach not feasible, as determined from the investigator assessment prior to docking the robot.
* Subject with adhesions, scarring and disease status in the body which in the opinion of the investigator limits the ability to perform the minimally invasive procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who will undergo the study specified procedure as primary procedure with da Vinci 5 robot and who meet all eligibility criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To assess the force imparted on the tissue by force feedback instruments. | Intra-operative

SECONDARY OUTCOMES:
To evaluate the utility of force feedback instruments during specific procedural steps or tasks. | Post-operative prior to discharge

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - St. David's Healthcare, Austin, Texas